CLINICAL TRIAL: NCT00001594
Title: Evaluation and Intervention for Ambulation, Growth, and Basilar Invagination in Osteogenesis Imperfecta
Brief Title: Evaluation and Intervention for the Effects of Osteogenesis Imperfecta
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970064; 97-CH-0064
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-07-23

CONDITIONS: Osteogenesis Imperfecta
Keywords: Natural History; Brittle Bone; Connective Tissue; Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with OI: Children with OI

SUMMARY:
We propose a longitudinal study of the natural history of types III and IV osteogenesis imperfecta for children age birth to 25 years. A consistent objective throughout this study is to obtain a comprehensive assessment of the natural history and progression of the multiple secondary features of osteogenesis imperfecta. In addition to radiographic, bone density, physical rehabilitation and dental manifestations, we will assess the cardiovascular, pulmonary, neurological, and audiology systems.

The major objectives of this protocol focus on rehabilitation and physical therapy studies, pulmonary and cardiovascular function, neurological features, audiological studies and genetic and molecular biology aspects of OI. A major objective in this study is to expand the intensive rehabilitation and physical therapy studies of children with types III and IV OI. This objective continues the work that has been done in the Rehabilitation Department of the Clinical Center for the past 20 years on these patients. However, the focus of this objective is changing to include studies of scoliosis and its effect on function, studies of chest proportions and rib deformities, and studies of nonkinetic variables related to motor performance, such as temperament, competence, coping, and resilience in children with OI. The second major objective is the longitudinal study of pulmonary function in children with types III and IV OI. It is well known that cardiopulmonary complications are a major cause of disability and death in adults with OI; the developmental patterns of these complications, and whether susceptible individuals can be identified in childhood, is unknown. The third major objective of these studies of secondary features is to determine the incidence of basilar invagination and develop a monitoring and management plan for this neurological feature. Next, the prevalence, severity, age of onset and genotypic/phenotypic correlation of hearing loss among children with types II and IV OI remains poorly understood; therefore, the study of audiological features is our fourth major objective. The final major objective in this study is the continued study of the genetic and molecular biology aspect of OI. Patients will have skin biopsies for collagen studies at the biochemical and molecular level. Parents will have blood drawn for determination of mosaic status for the mutation that causes their child s OI. These studies will provide further information on genotype/phenotype correlation and other variables in OI genetics. As appropriate, bone chips from emergency or elective surgical procedures on the participants will be used to study osteoblast function in OI.

DETAILED DESCRIPTION:
We propose a longitudinal study of the natural history of types III and IV osteogenesis imperfecta for children age birth to 30 years. A consistent objective throughout this study is to obtain a comprehensive assessment of the natural history and progression of the multiple secondary features of osteogenesis imperfecta. In addition to radiographic, bone density, physical rehabilitation and dental manifestations, we will assess the cardiovascular, pulmonary, neurological, and audiology systems.

The major objectives of this protocol focus on rehabilitation and physical therapy studies, pulmonary and cardiovascular function, neurological features, audiological studies and genetic and molecular biology aspects of OI. A major objective in this study is to expand the intensive rehabilitation and physical therapy studies of children with types III and IV OI. This objective continues the work that has been done in the Rehabilitation Department of the Clinical Center for the past 20 years on these patients. However, the focus of this objective is changing to include studies of scoliosis and its effect on function, studies of chest proportions and rib deformities, and studies of nonkinetic variables related to motor performance, such as temperament, competence, coping, and resilience in children with OI. The second major objective is the longitudinal study of pulmonary function in children with types III and IV OI. It is well known that cardiopulmonary complications are a major cause of disability and death in adults with OI; the developmental patterns of these complications, and whether susceptible individuals can be identified in childhood, is unknown. The third major objective of these studies of secondary features is to determine the incidence of basilar invagination and develop a monitoring and management plan for this neurological feature. Next, the prevalence, severity, age of onset and genotypic/phenotypic correlation of hearing loss among children with types II and IV OI remains poorly understood; therefore, the study of audiological features is our fourth major objective. The final major objective in this study is the continued study of the genetic and molecular biology aspect of OI. Patients will have skin biopsies for collagen studies at the biochemical and molecular level. Parents will have blood drawn for determination of mosaic status for the mutation that causes their child s OI. These studies will provide further information on genotype/phenotype correlation and other variables in OI genetics. As appropriate, bone chips from emergency or elective surgical procedures on the participants will be used to study osteoblast function in OI.

ELIGIBILITY:
* INCLUSION CRITERIA:

Children will be recruited from the United States. This recruitment will be accomplished by our contacts with the Osteogenesis Imperfecta Foundation, parent-to-parent communication, and outside referrals from other health care providers.

There are no exclusionary criteria related to race or gender for this protocol.

Children enrolled in this study will be limited to those with Sillence Types III and IV OI, as determined by clinical and genetic criteria.

Patients age birth to 10 years at enrollment will be considered for this protocol.

Children who have not had skin biopsy done for collagen analysis at another facility are preferred for participation in this study. However, previous skin biopsy at another facility will not preclude participation in this protocol.

EXCLUSION CRITERIA:

Children who can be expected to attain at least some degree of ambulatory skill or have high potential for achieving independent locomotion with assistive technology.

Children who are clinically too severe to benefit from this program are defined by the following criteria:

1. The ratio of head circumference age (the age for which the child's head or body size falls at the 50th percentile) to body length age (the age for which the child's length falls at the 50th percentile) is 7:1 or greater;
2. Children who are 24 months of age, and who are unable to sit unsupported for 60 seconds and are unable to demonstrate the ability to prop themselves on upper extremities in the prone position;
3. Children who have other significant medical problems, especially severe cardiopulmonary problems, which have an impact on their physical development.

Compliance with the visit schedule, maintenance of the physical therapy program, and completion of the measurement tools are central to our analysis of the outcomes of this study. Failure to comply with these conditions will constitute exclusion criteria.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children will be recruited from the United States. This recruitment will be accomplished by our contacts with the Osteogenesis Imperfecta Foundation, parent-to-parent communication, and outside referrals from other health care providers
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 1997-01-29 (Actual)

PRIMARY OUTCOMES:
Ambulation, Basilar Invagination, Secondary Effects of OI | age-based
  For the younger children, we evaluated bone density, physical function, dental manifestations, and the cardiovascular, pulmonary, and audiologic systems. Visits for children under 5 will be every 4 months. These assessments will continue when the participants turn 5, with the addition of the neurological system. All children ages 5-18 years will be evaluated at the Clinical Center every 6 months. Ages 19- will be seen on an annual basis

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Zimmerberg, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Due to the data in this natural history study being open and utilized in comparison with another currently open, longitudinal, natural history study, we would wait for that open study to meet its primary and secondary endpoints prior to making the plan to make IPD available.

REFERENCES:
- [Background] Marini JC. Osteogenesis imperfecta: comprehensive management. Adv Pediatr. 1988;35:391-426. No abstract available. PMID 3055864
- [Background] Marini JC, Bordenick S, Heavner G, Rose S, Hintz R, Rosenfeld R, Chrousos GP. The growth hormone and somatomedin axis in short children with osteogenesis imperfecta. J Clin Endocrinol Metab. 1993 Jan;76(1):251-6. doi: 10.1210/jcem.76.1.8421094.
- [Background] Charnas LR, Marini JC. Communicating hydrocephalus, basilar invagination, and other neurologic features in osteogenesis imperfecta. Neurology. 1993 Dec;43(12):2603-8. doi: 10.1212/wnl.43.12.2603. PMID 8255464
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-CH-0064.html